CLINICAL TRIAL: NCT00885547
Title: Prospective Clinical Study of TW in Treatment of IgAN With Asymptomatic Abnormal Urinalysis.
Brief Title: Prospective Study of TW in Treatment of IgAN With Asymptomatic Abnormal Urinalysis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low-rate of enrollment
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhi-Hong Liu, M.D., professor, Nanjing University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-0904
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- immunosuppressor (Experimental)
  Interventions: Drug: tripterygium wilfordii (TW)

INTERVENTIONS:
Drug: tripterygium wilfordii (TW) — 90 mg/d for 6 months
  Other Names: tripterygium wilfordii

SUMMARY:
The purpose of this study is to:

1. To evaluate the latest effects of TW for IgA nephropathy (IgAN) with asymptomatic abnormal urinalysis.
2. To evaluate the safety and tolerability of TW.

DETAILED DESCRIPTION:
Patients who fit the inclusion criteria will be randomly divided into three groups: TW group (TW at dosage of 90 mg/d), ARB group (the control group, valsartan at dosage of 160 mg/d) and combined treatment group (TW at dosage of 60 mg/d and valsartan at dosage of 80 mg/d).

ELIGIBILITY:
Inclusion Criteria:

1. 18-60 years old but no requirement for gender
2. All well fit the Diagnostic Criteria for Primary IgAN and IgAN with asymptomatic abnormal urinalysis
3. Informed consent is obtained from each research subject who agrees to conduct a periodic follow-up according to the research arrangement

Exclusion Criteria:

1. Secondary IgA nephropathy, such as Henoch-Schönlein purpura nephritis, Lupus nephritis and so on
2. Some secondary kidney diseases like diabetic nephropathy or other systemic diseases which may effect the pathologic and physiological function of kidney like hypertension and arteriosclerosis
3. Severe infection
4. Abnormality of liver function with glutamic pyruvic transaminase (GPT) or glutamic-oxal(o)acetic transaminase (GOT) more than twice upper limit of normal
5. Women during pregnancy and lactation
6. Patients need to procreation lately
7. Patients treated with TW or ARB within 4 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2009-03; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The percentage got to complete remission (CR) of TW group, the combined treatment group, and the control group after the 3, 6 months treatment. | 12 months

SECONDARY OUTCOMES:
The percentage of total effect of the 3 groups and adverse event within the follow-up periods. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Tang, Doctor, Principal Investigator — Nanjing University School of Medicine